CLINICAL TRIAL: NCT00296231
Title: Nasal High Frequency Ventilation in Preterm Infants: A Pilot Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tarah T Colaizy (Other)
Responsible Party: Sponsor-Investigator, Tarah T Colaizy, Associate Professor of Pediatrics, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 200508714
Record Dates: First submitted 2006-02-22; First posted 2006-02-24 (Estimated); Results first posted 2010-12-22 (Estimated); Last update posted 2018-02-09 (Actual); Status verified 2018-01

CONDITIONS: Infant Respiratory Distress Syndrome; Respiratory Insufficiency; Apnea of Prematurity
Keywords: premature infants; very low birthweight infants; high frequency ventilation; nasal ventilation
MeSH Terms: conditions — Pulmonary Atelectasis; Respiratory Insufficiency; Apnea; Premature Birth

ARMS (1):
- Nasal High Frequency Ventilation (Experimental): Stable infants born at less than 1501 g who are at least 7 days old and undergoing nasal continuous positive airway pressure treatment.
  Interventions: Other: Nasal high frequency ventilation

INTERVENTIONS:
Other: Nasal high frequency ventilation — use of the high frequency ventilation mode of the Infant Star ventilator via a single nasopharyngeal prong.

SUMMARY:
The purpose of this study is to test whether application of high frequency ventilation through a nasal tube can lower blood carbon dioxide levels in stable preterm infants.

DETAILED DESCRIPTION:
Prolonged mechanical ventilation is frequently needed to treat respiratory insufficiency and apnea in very low birthweight (VLBW, <1500 g) preterm infants. Endotracheal intubation and mechanical ventilation carry many risks including potentially fatal air leaks and ventilator-associated pneumonias. Less-invasive methods of respiratory support are needed to minimize these risks while supporting the convalescing preterm infant. We propose to test the effectiveness of nasal high-frequency ventilation (NHFV) in stable neonates with mild respiratory acidosis who are dependent on nasal continuous positive airway pressure for respiratory support (CPAP). Nasal high frequency ventilation may be effective in decreasing rates of reintubation for apnea or respiratory insufficiency in VLBW infants. We will enroll 60 stable VLBW infants who are currently being treated with nasal CPAP and who have mild respiratory acidosis. Twenty patients will be assigned to each ventilator under investigation. Nasal high frequency ventilation will be applied at the same mean airway pressure as the patients' previous CPAP support. The amplitude on nasal high frequency ventilation will be adjusted to achieve adequate shaking of the chest wall. Blood gas measurements, transcutaneous continuous pCO2 monitoring, continuous pulse oximetry, and chest x-rays will be used to assess safety and efficacy. Study power has been calculated to detect a difference (drop or rise) in partial pressure of CO2 (pCO2) equal to two-thirds of the standard deviation of pCO2 change reported in another study (van der Hoeven et al., 1998), which is a clinically relevant difference.

ELIGIBILITY:
Inclusion Criteria:

* birthweight less than 1500 g
* Age >7 days
* Free of severe intraventricular hemorrhage (Grade III-IV)
* requiring nasal continuous positive airway pressure with a stable compensated respiratory acidosis (pH 7.25 - 7.45, pCO2 > 43 mm Hg),
* medically stable.

Exclusion Criteria:

* major congenital anomalies

Ages: 7 Days to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2006-02; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tarah T Colaizy, MD, MPH, Principal Investigator — University of Iowa
Locations (1):
- Children's Hospital of Iowa NICU, Iowa City, Iowa, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Nassal High Frequency Ventilation: Stable infants, born at less than 1501 g birthweight, who were at least 7 days of age and requiring nasal continuous positive airway pressure ventilatory support
Period: Overall Study
Arm/Group | Nassal High Frequency Ventilation
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Nassal High Frequency Ventilation
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: days] | 39.5 [18 to 147]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: pCO2 Measurements Post-intervention, as Compared to Pre-intervention Values
Description: Capillary partial pressure of CO2 (pCO2) was measured before and after 2 hours of nasal high frequency ventilatiion in a group of subjects. Each served as his/her own control.
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nassal High Frequency Ventilation
Number analyzed (Participants) | 14
mm Hg
  pre-nasal high frequency ventilation pCO2 | 50 (6)
  post-nasal high frequency ventilation pCO2 | 45 (9)
Statistical Analysis 1: Comparison: Nassal High Frequency Ventilation; Paired Student's t-test was used to compare pre and post intervention pCO2 values; Test type: Superiority or Other; p = 0.011, t-test, 2 sided

2. Secondary Outcome: Transcutaneous CO2 Measurements as a Trend Throughout Intervention
Description: We used a transcutaneous CO2 monitor (TCOM) as a safety device throughout the study. We analyzed the change in TCOM readings recorded every 30 minutes (5 measurements) to determine safety
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: torr
Arm/Group | Nassal High Frequency Ventilation
Number analyzed (Participants) | 14
torr
  pre-nasal high frequency TCOM | 47 (5)
  post-nasal high frequency ventilation TCOM | 46 (5)

ADVERSE EVENTS:
Arm/Group | Nassal High Frequency Ventilation
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes